CLINICAL TRIAL: NCT04138498
Title: A Randomized, Single-dose, Four-sequence, Four-period, Crossover Study in Adult ADHD Subjects to Establish Safety, Tolerability, and Comparative Bioavailability of CTx-1301 (Dexmethylphenidate) to Focalin XR™ Under Fasted Conditions
Brief Title: CTx-1301 Comparative Bioavailability Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cingulate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CTx-1301-001
Record Dates: First submitted 2019-09-19; First posted 2019-10-24 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: ADHD
Keywords: ADHD; bioavailability; dexmethylphenidate; BA study; dMPH; d-MPH
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride; Capsules; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (ADBC) (Experimental): Subjects in sequence ADBC will receive study treatments in the following order: Focalin XR 5 mg capsule, CTx-1301 50 mg tablet, CTx-1301 6.25 mg tablet, Focalin XR 40 mg capsule.
  Interventions: Drug: Dexmethylphenidate 5 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 6.25 mg Tablet; Drug: Dexmethylphenidate 40 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 50 mg Tablet
- Sequence 2 (BACD) (Experimental): Subjects in sequence BACD will receive study treatments in the following order: CTx-1301 6.25 mg tablet, Focalin XR 5 mg capsule, Focalin XR 40 mg capsule, CTx-1301 50 mg tablet.
  Interventions: Drug: Dexmethylphenidate 5 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 6.25 mg Tablet; Drug: Dexmethylphenidate 40 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 50 mg Tablet
- Sequence 3 (CBDA) (Experimental): Subjects in sequence CBDA will receive study treatments in the following order: Focalin XR 40 mg capsule, CTx-1301 6.25 mg tablet, CTx-1301 50 mg tablet, Focalin XR 5 mg capsule.
  Interventions: Drug: Dexmethylphenidate 5 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 6.25 mg Tablet; Drug: Dexmethylphenidate 40 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 50 mg Tablet
- Sequence 4 (DCAB) (Experimental): Subjects in sequence DCAB will receive study treatments in the following order: CTx-1301 50 mg tablet, Focalin XR 40 mg capsule, Focalin XR 5 mg capsule, CTx-1301 6.25 mg tablet.
  Interventions: Drug: Dexmethylphenidate 5 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 6.25 mg Tablet; Drug: Dexmethylphenidate 40 Mg Oral Capsule, Extended Release; Drug: Dexmethylphenidate 50 mg Tablet

INTERVENTIONS:
Drug: Dexmethylphenidate 5 Mg Oral Capsule, Extended Release — Reference listed drug (RLD) for comparative BA evaluation
  Other Names: Focalin XR (dexmethylphenidate) 5 mg Capsule
Drug: Dexmethylphenidate 6.25 mg Tablet — Experimental drug for comparative BA evaluation
  Other Names: CTx-1301 (dexmethylphenidate) 6.25 mg Tablet
Drug: Dexmethylphenidate 40 Mg Oral Capsule, Extended Release — Reference listed drug (RLD) for comparative BA evaluation
  Other Names: Focalin XR (dexmethylphenidate) 40 mg capsule
Drug: Dexmethylphenidate 50 mg Tablet — Experimental drug for comparative BA evaluation
  Other Names: CTx-1301 (dexmethylphenidate) 50 mg tablet

SUMMARY:
The primary purpose of this study is to compare the bioavailability of CTx-1301 (dexmethylphenidate) to the registered listed drug, Focalin XR and to evaluate dose proportionality of CTx-1301. In addition, this study seeks to characterize the pharmacokinetics of dexmethylphenidate and evaluate the safety and tolerability of CTx-1301.

DETAILED DESCRIPTION:
The study will comprise of a randomized, single-dose, four-sequence, four-period, in-clinic crossover study in approximately 36 adult ADHD subjects. All subjects considered eligible at Screening will proceed to tolerability test day, dosing 40 mg Focalin XR to evaluate safety and tolerability of the higher dose of d-MPH. If subject is able to safely tolerate the test dose, and meets all inclusion/exclusion criteria, they will be considered eligible for randomization into the study. All subjects will be randomized to receive four treatments throughout the course of the study; one CTx-1301 trimodal d-MPH tablet containing 6.25 mg d-MPH, one Focalin 5 mg XR capsule, one CTx-1301 50 mg tablet, and one 40 mg Focalin XR capsule. Administration of study drug will occur only on Assessment Days; no study drug will be administered during screening or unscheduled days (USVs).

The lowest and highest doses of CTx-1301 (dexmethylphenidate, 6.25 and 50 mg) were selected to bridge to the lowest and highest doses of Focalin XR (dexmethylphenidate, 5 and 40 mg) in this comparative BA study.

ELIGIBILITY:
Inclusion Criteria:

1. Gender

   a. Male or Female
2. Age

   a. Aged between 18 and 55 years inclusive.
3. Weight and BMI

   1. Body weight ≥ 50 kg
   2. BMI ≥ 18 and ≤ 35
4. Compliance

   1. Understands and is willing, able and likely to comply with all study procedures and restrictions.
   2. If sexually active, male subjects must use the double-barrier method (condom and spermicide) for birth control during the study and for 90 days following the last administration of study drug.
   3. If sexually active, female subjects of child-bearing potential must use an acceptable method of contraception, including abstinence from heterosexual intercourse, hormonal contraceptives, intrauterine device (IUD) with or without hormones, or double-barrier method (e.g. condom and spermicide), during the study and for 30 days following the last administration of study drug.
   4. Male subjects must agree not to donate sperm during the study and for 90 days following the last administration of study drug.
   5. Female subjects must agree not to donate eggs during the study and for 30 days following the last administration of study drug.
5. Consent a. Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent (signed and dated) obtained before any study-related activities are performed.
6. Indication

   1. Subject must report history of diagnosis of ADHD.
   2. If subject is currently taking stimulant medication, they must be willing and able to safely abstain from any other ADHD treatment during 96 hrs. prior to check-in on Day -4 and through the complete duration of the study.
7. General Health

   1. Good general health (in the opinion of an investigator) with no clinically significant or relevant abnormalities on medical history or physical examination which could affect the safety of the subject or study data.
   2. No vomiting or fever within 24-hours of check-in at Day -4
   3. Subject has sufficient venous access to allow cannulation and/or venipuncture to obtain the required volume of blood for this study.
   4. Subject must currently be taking or previously have taken a stimulant medication for ADHD.
8. Smoking/Caffeine/Alcohol

   1. Subject must be able to refrain from smoking cigarettes 1 hour prior to dosing and 7 hours after dosing on dosing days. Subject must agree not to smoke more than one cigarette per hour, not to exceed 10 cigarettes per day.
   2. Subject must be able to refrain from caffeine for 10 hours prior to check-in at Day -4 and for the duration of the study.
   3. Subject must be able to refrain from using alcohol 48 hrs. prior to Day -4 and for the duration of the study.
9. ADHD Medication History

   1. Subject's medication history suggests they will be able to tolerate a 40 mg dose of dexmethylphenidate.
   2. Subject must demonstrate tolerability of dexmethylphenidate assessed by tolerability day/test dose of 40 mg Focalin XR as evaluated by the investigator.

Exclusion Criteria:

1. Medical History

   1. Current and/or recurrent disease or illness that, in the opinion of an investigator, could affect the study conduct, study outcome, subject safety, or pharmacokinetic (PK) assessments (e.g., hepatic disorders, renal insufficiency, non-self-limiting gastrointestinal disorders, congestive heart failure).
   2. Current and/or previous history of any other serious, severe or unstable psychiatric illness which in the opinion of the investigator, may require treatment (e.g. anxiety, psychosis, mood disorder, motor tics or suicidality) or make the subject unlikely to fully complete the study, and/or any condition that presents undue risk from the study medication or procedures.
   3. Subject cannot have suicidal thoughts within the last 6 months as supported by the Columbia Suicide Severity Rating Scale (C-SSRS).
   4. Positive test results for Human Immunodeficiency Virus (HIV)-1/HIV-2 antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibody (HCVAb).
   5. A family history of sudden cardiac or unexplained death.
   6. Any condition or abnormal laboratory finding that could result in harm to the subject, affect the outcome of the study, or suggest unstable medical illness.
   7. As a result of the MINI, medical history, physical examination, and/or screening investigations (including ECG results, vital signs and/or laboratory abnormality), an Investigator considers the subject disqualified for the study.
   8. Subject plans to undergo elective procedures/surgery at any time during the study.
   9. Subject has had surgery within the past 90 days.
   10. Subject of child-bearing potential is pregnant or planning to become pregnant during the duration of the study or within 30 days of the end of the study.
   11. Subject is breast-feeding during the study or within 30 days of the study.
2. Medications

   a. Subject has taken any medication that, in the opinion of an Investigator, has been shown to alter the PK of d-MPH.

   b. Use of any prescription medication within 14 days prior to Day -3 (ADHD medications must be discontinued at least 96 hours prior to check-in at Day -4), and/or use of any OTC medications (such as antacids, vitamins, minerals, dietary/herbal preparations, and nutritional supplements) within 7 days prior to Day -3 unless jointly approved by an Investigator and Sponsor.

   i. Subjects are permitted to take hormonal contraceptives and hormone replacement therapy at acceptable levels if stable at least 30 days prior to Day -4, through the duration of the study, and for 30 days after the study ends.

   ii. Acetaminophen (up to 2 grams per day) may be used during the study under the direction of the Investigator.

   iii. On a case-by-case basis, an Investigator is permitted to allow the use of certain concomitant medications, for example, to treat an AE, as long as an Investigator determines that the medication will not affect the subject's safety or study integrity (eg, topical medications).
3. Alcohol/Substance Abuse

   1. Recent history (within the last year) of alcohol or other substance abuse.
   2. Subject has positive breath alcohol test or urine test for drugs of abuse at screening or check-in (prescribed ADHD medication is acceptable during screening but must be stopped at least 96 hrs prior to check in at Day -4). Note: At the discretion of an Investigator, the tests may be repeated. If THC is positive at screening or check-in, a cannabis intoxication evaluation will be done by an investigator at check-in only; inclusion will be at the investigator's discretion, due to the slow release of THC from adipose tissue.
4. Smoking

   a. Subject regularly smokes more than 10 cigarettes/day (or other nicotine-containing products) or Subject has recently discontinued smoking (within the last 3 months)
5. Allergy/Intolerance

   a. Subject has a history of allergy to d-MPH, to any component of the dosage form, or any other allergy, which, in the opinion of an Investigator, contraindicates their participation.
6. Clinical Studies

   1. Participation in another investigational product study (inclusive of final post-study examination) or receipt of an investigational drug within the 30 days before screening day.
   2. Previous participation in this study.
7. Personnel

   a. An employee of the sponsor, study site, or members of their immediate family.
8. Blood

   1. Subject has donated blood, plasma, or experienced significant blood loss (excess of 500 ml) within 3 months of screening and for the duration of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Brams, MD, Study Director — Sponsor Medical Officer
Locations (1):
- Vince & Associates, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at a single site from November 22, 2019 to March 06, 2020.
Pre-assignment Details: Of 106 subjects who were screened, 45 (42.5%) were enrolled into the study and randomized to a sequence of treatment.
Groups:
- Sequence 1 (ADBC): Subjects in sequence ADBC received study treatments in the following order: Focalin XR 5 mg capsule, CTx-1301 50 mg tablet, CTx-1301 6.25 mg tablet, Focalin XR 40 mg capsule.
  Dexmethylphenidate 5 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 6.25 mg Tablet: Experimental drug for comparative BA evaluation
  Dexmethylphenidate 40 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 50 mg Tablet: Experimental drug for comparative BA evaluation
- Sequence 2 (BACD): Subjects in sequence BACD received study treatments in the following order: CTx-1301 6.25 mg tablet, Focalin XR 5 mg capsule, Focalin XR 40 mg capsule, CTx-1301 50 mg tablet.
  Dexmethylphenidate 5 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 6.25 mg Tablet: Experimental drug for comparative BA evaluation
  Dexmethylphenidate 40 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 50 mg Tablet: Experimental drug for comparative BA evaluation
- Sequence 3 (CBDA): Subjects in sequence CBDA received study treatments in the following order: Focalin XR 40 mg capsule, CTx-1301 6.25 mg tablet, CTx-1301 50 mg tablet, Focalin XR 5 mg capsule.
  Dexmethylphenidate 5 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 6.25 mg Tablet: Experimental drug for comparative BA evaluation
  Dexmethylphenidate 40 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 50 mg Tablet: Experimental drug for comparative BA evaluation
- Sequence 4 (DCAB): Subjects in sequence DCAB received study treatments in the following order: CTx-1301 50 mg tablet, Focalin XR 40 mg capsule, Focalin XR 5 mg capsule, CTx-1301 6.25 mg tablet.
  Dexmethylphenidate 5 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 6.25 mg Tablet: Experimental drug for comparative BA evaluation
  Dexmethylphenidate 40 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
  Dexmethylphenidate 50 mg Tablet: Experimental drug for comparative BA evaluation
Period: Overall Study
Arm/Group | Sequence 1 (ADBC) | Sequence 2 (BACD) | Sequence 3 (CBDA) | Sequence 4 (DCAB)
Started | 11 | 10 | 12 | 12
Completed | 10 | 10 | 10 | 9
Not Completed | 1 | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (ADBC) | Sequence 2 (BACD) | Sequence 3 (CBDA) | Sequence 4 (DCAB) | Total
Number analyzed (Participants) | 11 | 10 | 12 | 12 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 12 | 12 | 45
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 5
  Male | 11 | 8 | 11 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 3 | 5
  Not Hispanic or Latino | 11 | 10 | 10 | 9 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 6 | 5 | 18
  White | 7 | 6 | 6 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 12 | 12 | 45
History of ADHD [Number; unit: participants] | 11 | 10 | 12 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: d-MPH Plasma concentration
Time Frame: Hours 0 to 28
Population: PK Completer Population
Measure: Geometric Mean (90% Confidence Interval); unit: pg/mL
Groups:
- Treatment A: Focalin XR 5 mg capsule
  Dexmethylphenidate 5 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
- Treatment B: CTx-1301 6.25 mg tablet
  Dexmethylphenidate 6.25 Mg Oral Tablet, Extended Release: Investigational Medication for comparative BA evaluation
- Treatment B/A: PK Comparison of 6.25 mg CTx-1301 (treatment B) to 5 mg Focalin XR (treatment A)
- Treatment C: Focalin XR 40 mg capsule
  Dexmethylphenidate 40 Mg Oral Capsule, Extended Release: Reference listed drug (RLD) for comparative BA evaluation
- Treatment D: CTx-1301 50 mg tablet
  Dexmethylphenidate 50 Mg Oral Tablet, Extended Release: Investigational Medication for comparative BA evaluation
- Treatment D/C: PK Comparison of 50 mg CTx-1301 (treatment D) to 40 mg Focalin XR (treatment C).
Arm/Group | Treatment A | Treatment B | Treatment B/A | Treatment C | Treatment D | Treatment D/C
Number analyzed (Participants) | 41 | 39 | 39 | 43 | 42 | 42
pg/mL | 3138.41 [2893.862 to 3403.633] | 2874.52 [2646.813 to 3121.816] | 0.92 [0.843 to 0.995] | 23884.13 [22050.942 to 25869.722] | 24685.37 [22774.231 to 26756.894] | 1.03 [0.953 to 1.120]

2. Primary Outcome: AUC(0-infinity)
Description: Area under the curve from time 0 extrapolated to infinite time
Time Frame: Hours 0 to 28
Population: PK Completer Population
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment B/A | Treatment C | Treatment D | Treatment D/C
Number analyzed (Participants) | 41 | 39 | 39 | 43 | 42 | 42
ng/mL | 24384.31 [22579.167 to 26333.776] | 27661.46 [25603.455 to 29884.885] | 1.13 [1.090 to 1.181] | 203127.64 [188123.507 to 219328.465] | 239317.53 [221590.471 to 258462.729] | 1.18 [1.133 to 1.225]

3. Primary Outcome: AUC(Last)
Description: AUC from time 0 to the last measurable concentration
Time Frame: Hours 0 to 28
Population: PK Completer Population
Measure: Geometric Mean (90% Confidence Interval); unit: pg/mL
Arm/Group | Treatment A | Treatment B | Treatment B/A | Treatment C | Treatment D | Treatment D/C
Number analyzed (Participants) | 41 | 39 | 39 | 43 | 42 | 42
pg/mL | 22793.45 [20666.366 to 25139.474] | 25540.99 [23149.418 to 28179.632] | 1.12 [1.075 to 1.169] | 190456.27 [172736.598 to 209993.654] | 221949.48 [201261.408 to 244764.129] | 1.17 [1.118 to 1.214]

4. Secondary Outcome: Partial AUCs
Description: AUC from Hours 0-3, 3-6, 6-9, 9-12, and 12 to 16
Time Frame: Hours 0 to 28
Measure: Geometric Mean (90% Confidence Interval); unit: hr*pg/mL
Arm/Group | Treatment A | Treatment B | Treatment B/A | Treatment C | Treatment D | Treatment D/C
Number analyzed (Participants) | 41 | 39 | 39 | 43 | 42 | 42
hr*pg/mL
  AUC0-3 | 4928.24 [4520.066 to 5373.276] | 3943.21 [3612.595 to 4304.075] | .80 [0.743 to 0.861] | 37963.37 [34854.010 to 41350.112] | 32744.35 [30044.791 to 35686.470] | .86 [0.803 to 0.927]
  AUC3-6 | 6939.76 [6357.221 to 7575.675] | 6317.47 [5778.203 to 6907.071] | 0.91 [0.831 to 0.997] | 51204.34 [46939.593 to 55856.559] | 51368.60 [47085.223 to 56041.632] | 1.00 [0.918 to 1.096]
  AUC6-9 | 5644.67 [5176.704 to 6154.948] | 5624.50 [5149.945 to 6142.780] | 1.00 [0.909 to 1.093] | 49159.01 [45116.976 to 53563.164] | 53313.02 [48889.077 to 58137.277] | 1.08 [0.991 to 1.187]
  AUC9-12 | 2769.68 [2498.675 to 3070.079] | 3638.05 [3277.387 to 4038.399] | 1.31 [1.198 to 1.440] | 25193.87 [22743.535 to 27908.203] | 34316.26 [30955.023 to 38042.466] | 1.36 [1.245 to 1.490]
  AUC12-16 | 1643.22 [1458.189 to 1851.741] | 3092.55 [2739.223 to 3491.455] | 1.88 [1.679 to 2.109] | 15739.33 [13978.890 to 17721.462] | 26183.15 [23231.791 to 29509.457] | 1.66 [1.488 to 1.860]

5. Secondary Outcome: K
Description: Rate at which a drug is removed from the system
Time Frame: Hours 0 to 28
Population: PK Completer Population
Measure: Geometric Mean (Standard Deviation); unit: (1/hr)
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 41 | 39 | 43 | 42
(1/hr) | 0.18 (0.053) | 0.16 (0.040) | 0.17 (0.035) | 0.16 (0.034)

6. Secondary Outcome: Half-life
Description: Time (Hours) it takes for the concentration of the drug in plasma to be reduced by 50%
Time Frame: Hours 0 to 28
Measure: Geometric Mean (Standard Deviation); unit: hr*pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 41 | 39 | 43 | 42
hr*pg/mL | 3.77 (1.066) | 4.32 (1.866) | 4.05 (0.977) | 4.21 (1.163)

7. Secondary Outcome: Tmax
Description: Time (Hours) after administration of a drug when the maximum plasma concentration is reached
Time Frame: Hours 0 to 28
Measure: Median (Full Range); unit: hr*pg/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 41 | 39 | 43 | 42
hr*pg/mL | 5.00 [1.0 to 7.0] | 5.00 [1.0 to 7.0] | 6.00 [1.0 to 8.0] | 5.00 [1.0 to 10.0]

8. Secondary Outcome: Tlag
Description: Delay (hours) between the time of dosing and time of appearance of concentration in the sampling
Time Frame: Hours 0 to 28
Population: PK Completer Population
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 41 | 39 | 43 | 42
hr | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.5]

9. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: TEAEs will be measured from Day 0 to Day 10 (End of Study)
Time Frame: Day 0 to Day 10
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 41 | 39 | 43 | 42
participants | 7 | 4 | 22 | 14

ADVERSE EVENTS:
Time Frame: Day -4 to Day 10
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 7/41 | 4/39 | 22/43 | 14/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=41) | Treatment B (N=39) | Treatment C (N=43) | Treatment D (N=42)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling Abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-Existing Condition Improved (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Change in Sustained Attention (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Frustration tolerance decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/PI shall not have the right to use the results pertaining to Institution's/PI's activities for their own instructional or research publication objectives, unless provided written permission by Sponsor. Publication must not disclose Confidential Information. Institution and PI shall submit in writing to Sponsor review of any Publication. Sponsor shall advise Institution of information which is Confidential Information or which may impair Sponsor's ability to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT04138498/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT04138498/SAP_001.pdf